CLINICAL TRIAL: NCT01623804
Title: Can Very Low Intensity Ultrasound Therapy Improve Pain in People With Knee Osteoarthritis? A Pilot Randomized Controlled Trial
Brief Title: Randomized Trial in knEe Osteoarthritis Using Low Intensity Ultrasound - Evaluating Feasibility (RELIEF)
Acronym: RELIEF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding to support alternate feasible recruitment strategy was not acquired
Sponsor: McMaster University (Other)
Collaborators: Bioventus LLC (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EX-KOA-1206; EX-KOA-xxxxxx (Other Grant/Funding Number: Smith & Nephew, Inc); MTP 108229/MTO 108232 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2012-05-31; First posted 2012-06-20 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Knee Osteoarthritis
Keywords: Ultrasound therapy; Tibiofemoral joint, medial; Nonsurgical
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low intensity, pulsed ultrasound (Active Comparator)
  Interventions: Device: low intensity, pulsed ultrasound
- Sham ultrasound (Sham Comparator)
  Interventions: Device: sham ultrasound

INTERVENTIONS:
Device: low intensity, pulsed ultrasound — 1.5MHz, spatial average-temporal average intensity = 0.03W/cm2, pulsed (burst frequency 1kHz, burst duration 200µm, duty cycle 20%); self-administered to the medial side of the knee joint while sitting down for 20 minutes every day for 3 months.
  Other Names: Exogen Express Ultrasound Bone Healing System
  Arms: Low intensity, pulsed ultrasound
Device: sham ultrasound — no ultrasonic energy emitted; self-administered to the medial side of the knee joint while sitting down for 20 minutes every day for 3 months
  Other Names: sham Exogen Express Ultrasound Bone Healing System
  Arms: Sham ultrasound

SUMMARY:
The purpose of this pilot study is to determine the feasibility of conducting a high quality clinical trial to investigate the effects of low intensity, pulsed ultrasound on knee osteoarthritis pain and physical function.

ELIGIBILITY:
Inclusion Criteria:

* over 40 years of age;
* have medial tibiofemoral compartment knee OA;
* have mild to moderate medial compartment radiographic OA severity (determined by the attending surgeon and/or Advanced Practice Physiotherapist on the basis of a standing x-ray or MRI scan depending upon which is available at initial consult);
* have stable ('not getting worse or better overall despite short-term fluctuations during the past three months') pain having an average intensity ≥ 3 and ≤ 8 on an 11-point verbal numeric rating scale, VNRS) in one knee which is aggravated by activity and eased with rest;
* limited pain from other lower extremity joints; and
* no change in first line pain medication in the past 2 months and willingness to forego alterations in pain medication for the duration of the study unless deemed medically necessary.

Exclusion Criteria:

* history of traumatic OA or previous surgical intervention in the knee or knee effusion;
* intra-articular injection of the knee in the previous 6 months;
* received ultrasound treatment for knee OA within the past 6 months;
* body weight changed ≥ 5% in the past 2 months;
* level of physical function insufficient to perform the required assessments or administer the intervention (e.g. intermittent claudication, severe peripheral neuropathy, active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, chronic pain, arthritis in joints other than the study knee, bone fracture in the past 3 months);
* conditions listed as precautions or unknown safety risks for using the EXOGEN EXPRESS ultrasound device (pregnant or nursing women, individuals with thrombophlebitis, vascular insufficiency, abnormal skin sensitivity, sensory paralysis, open wound at the medial joint line of the knee, taking steroids/anti-coagulants, prescription non-steroidal anti-inflammatory, calcium channel blocker or applying the EXOGEN EXPRESS in close proximity to someone wearing a cardiac pacemaker);
* unable to read, write and/or understand English;
* other illness or reasons judged by the participant, clinicians or researchers to make participation inadvisable (e.g. plans to move or travel, cognitive deficit resulting in difficulty comprehending and complying with instructions, caregiving demands/lack of social support for participation);
* unwillingness to sign informed consent; or
* participation in a competing study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Rate of recruitment | 6 months
  Ability to recruit 30 participants over a 6 month period
Adherence to study protocol | 26 weeks
  Percent adherence to the protocols for randomization, recruitment, intervention, and assessment
Rate of retention | 26 weeks
  Number of participants completing the trial
Rate of all adverse events | 26 weeks
  Participants will be asked about serious and non-serious adverse events weekly during the 13 week intervention phase and monthly during the 13 week follow up phase. All adverse events will be recorded and addressed as indicated.

SECONDARY OUTCOMES:
Western Ontario and McMaster Osteoarthritis Index (WOMAC)3.1NPR pain subscale | 13 weeks
  Change from baseline in pain at 13 weeks
Western Ontario and McMaster Osteoarthritis Index (WOMAC)3.1NPR physical function subscale | 26 weeks
  Change from baseline in Physical Function at 26 weeks
6 Minute Walk Test (6MWT) | 26 weeks
  Change from baseline distance (metres) walked in 6 minutes at 26 weeks
SF-36 (RAND 36-item Health Survey 1.0) | 26 weeks
  Change from baseline in Health Related Quality of Life at 26 weeks
Global Rating of Disease Severity | 26 weeks
  Change from baseline in Global Rating of Disease Severity at 13 and 26 weeks will be assessed using an 11-point scale ('Considering all the ways that your knee arthritis affects you, please rate how you are doing on a scale from 0 (very well) to 10 (very poor))
11-point Verbal Numeric Rating Scale (VNRS) | 0 and 13 weeks
  Change from baseline in pain intensity (average, minimum and maximum over the past 24 hours and following physical performance tests)
Lower Extremity Functional Scale (LEFS) | 26 weeks
  Change from baseline in physical function at 26 weeks
Stair Climb test | 26 weeks
  Time (seconds) to ascend and descend a staircase with 9 steps
Perceived change | 13 and 26 weeks
  Perceived change from baseline will be assessed at 13 and 26 weeks using an 11-point scale ('With respect to your OA knee treated with ultrasound, how would you describe yourself now compared to baseline assessment?' -5 = a very great deal worse, 0 = about the same, +5 = a very great deal better)

CONTACTS AND LOCATIONS:
Overall Officials: Norma J MacIntyre, PT, PhD, Principal Investigator — McMaster University
Locations (1):
- Regional Joint Assessment Program - HHS/SJHH, Hamilton, Ontario, Canada